CLINICAL TRIAL: NCT01128673
Title: MRI Thermal Imaging of Infants Undergoing Cooling for HIE
Brief Title: MRI Thermal Imaging of Infants Undergoing Cooling for Hypoxic Ischemic Encephalopathy(HIE)
Status: Withdrawn | Type: Observational
Why Stopped: No funding
Sponsor: Vanderbilt University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, William Walsh, Chief of Nurseries, Vanderbilt University
Other Study IDs: 090575Walsh; NCT00993564 (obsolete NCT alias)
Record Dates: First submitted 2010-05-20; First posted 2010-05-24 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Hypoxic Ischemic Encephalopathy
Keywords: Hypoxic Ischemic encephalopathy; Magnet resonance imaging; Selective Head cooling; Therapeutic hypothermia
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Body Cooled: Infants undergoing total body cooling for HIE
  Interventions: Device: mRI
- HIE,Selective Head Cooled: Infants undergoing head cooling for HIE
  Interventions: Device: mRI

INTERVENTIONS:
Device: mRI

SUMMARY:
Hundreds of babies in the world are being treated with brain cooling to prevent brain injury after they lose oxygen at birth. This study will use the newly developed information from the magnet resonance image to determine the actual temperature of the brain. This will enable us to determine if the brain is being uniformly cooled and if techniques that provide cooling need to be changed to improve the injury prevention from cooling.

DETAILED DESCRIPTION:
We propose to develop a non-invasive measurement of brain tissue temperature and to apply this measurement of infants under-going cooling for HIE

1. We propose to do this by refining the use of the MRI evaluation of the NAA-H20 frequency shift. This molecular relationship is quite accurate (based on preliminary studies of an NAA-H20 phantom subject to controlled temperature variations) for measuring relative temperature changes.
2. The next step will be to perform further phantom imaging with continuous temperature measurements and to expand the phantom model. This work needs funding support to be completed.
3. At the same time we will be applying the MRI thermal imaging protocol to infants whom have experienced HIE and who are being treated with hypothermia to ameliorate the HIE. We have IRB approval to approach families and to obtain the required data during clinically indicated MRI scans, this data accumulation will add an additional 3-5 minutes to the MRI. We will then perform a second MRI after the infant is rewarmed. We will compare the pairs of readings at two different core temperatures from at least five regions of the brain.
4. We will evaluate results of regional temperature measurements to determine if cooling of the human infant brain is uniform.
5. We will compare the two modalities of cooling to determine if selective head cooling and total body cooling provide similar distribution of cooling.
6. The final goal will be to compare MRI identified injury patterns to the temperature distribution in order to determine if distribution of cooling is related to outcome.

ELIGIBILITY:
Inclusion Criteria:

* Infants in the NICU who are treated with hypothermia for hypoxic ischemic encephalopathy and who are scheduled to have an MRI for evaluation of the extent of their injury.
* Parent and attending physician consent to perform evaluation of MRI thermography.

Exclusion Criteria:

* Infants too unstable to have MRI scan, defined by being on any cardiac pressor medications or more than 40% oxygen on the ventilator.
* Infants too active to obtain MRI without sedation.

Max Age: 1 Week | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants with Hypoxic ischemic encephalopathy undergoing cooling
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2018-05 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Brain temperature | Day three of cooling
  MRI data will be used to estimate regional brain temperature

SECONDARY OUTCOMES:
Brain temperature upon rewarming | 2 hours after initial MRI
  Estimate of brain temperature when rewarmed

CONTACTS AND LOCATIONS:
Locations (1):
- Monroe Carell Jr Children's Hospital at Vanderbilt, Nashville, Tennessee, United States

REFERENCES:
- [Background] Magnetic Resonance Thermal Imaging 5th International Conference on Brain Monitoring and Imaging William F. Walsh1, Jason E. Moore3,4, Subechhya Pradhan3,4, Curtis Wuschensky2, J. Christopher Gatenby3,5, E. Brian Welch3,6 1Division of Neonatology, Vanderbilt University Medical Center, Nashville, TN 2Neuroradiology, Vanderbilt University Medical Center, Nashville, TN 3Institute of Imaging Science, Vanderbilt University, Nashville, TN 4Department of Physics and Astronomy, Vanderbilt University, Nashville, TN 5Department of Biomedical Engineering, Vanderbilt University, Nashville, TN 6Philips Healthcare, Cleveland, OH